CLINICAL TRIAL: NCT03877380
Title: Identification of Difficulties During a First Request for a Personal Autonomy Allowance by Beneficiaries and Identification of the Role of the Attending Physician During This Request.
Brief Title: Identification of Difficulties During a First Request for a Personal Autonomy Allowance
Acronym: IDAPA
Status: Completed | Type: Observational
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 35RC18_3040_IDAPA
Record Dates: First submitted 2019-01-30; First posted 2019-03-15 (Actual); Last update posted 2019-03-22 (Actual); Status verified 2019-03

CONDITIONS: Persons Requesting a Resource Allocation (APA); Beneficiairies Requesting a Resource Allocation (APA)
Keywords: personalised autonomy allowance; difficulties; physician's role

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: semi-structured interview — Semi-strucured interview to identify the difficulties when first applying for a personalised autonomy allowance by beneficiaries and their relatives

SUMMARY:
The objective of this study is to identify the difficulties when first applying for a first Resource Allocation (Personal autonomy allowance - APA) by beneficiaries and their relatives through a qualitative study and secondarily identification of the role of the attending physician during this request.

DETAILED DESCRIPTION:
The APA, introduced since the French law of 2001 aims to improve the care of people with loss of autonomy.

A regular assessment of autonomy in the elderly should be carried out in order to implement ABS as early as possible. The aim is to set up the necessary home help to avoid or delay institutionalisation.

It therefore seems essential to place oneself on the side of the beneficiaries and their relatives in order to identify the difficulties encountered during a first ABS application and their expectations as to the role of the general practitioner during this application?

ELIGIBILITY:
Inclusion Criteria:

* Beneficiaries living in Ille et Vilaine
* requesting for the first time a Resource Allocation (APA)

Or

* Persons requesting for the first time a Resource Allocation (APA)
* Allocation of resources for the benefit of a person residing in Ille et Vilaine

Exclusion Criteria:

* Refusal of Resource Allocation
* opposition to participation in the survey.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The population studied includes all the people who apply for a first Resource Allocation (APA) in all 6 territories of the department of Ille et Vilaine
Sampling Method: Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2018-06-13 (Actual); Primary Completion 2018-11-15 (Actual); Study Completion 2018-11-15 (Actual)

PRIMARY OUTCOMES:
Semi-structured interview | through study completion, an average of 1 year
  The interview guide will seek to make the beneficiaries talk about their administrative difficulties, access to information, coordination between medical and social professionals and others faced when making their first request for resource allocation (APA)

CONTACTS AND LOCATIONS:
Overall Officials: Emilie MENAND, MD, Principal Investigator — Rennes University Hospital
Locations (1):
- Conseil Départemental -Pôle Solidarité Humaine, Rennes, France